CLINICAL TRIAL: NCT05176938
Title: Effect of Preoperative Ultrasound Guided Thoracic Interfascial Plane Block Versus Preoperative Thoracic Erector Spinae Plane Block on Acute and Chronic Pain After Modified Radical Mastectomy
Brief Title: Effect of Ultrasound Guided Thoracic Interfascial Plane Block Versus Erector Spinae Plane Block After Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Areeg Kotb Ghalwash, Assistant lecturer of Anesthesiology and Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 33645/1/20
Record Dates: First submitted 2021-11-22; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Pain, Acute; Erector Spinae Plane Block; Mastectomy, Modified Radical; Thoracic Interfascial Plane Block; Pain, Chronic
MeSH Terms: conditions — Acute Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasound guided Thoracic Interfascial plane Block (TIFB) (Experimental): Patients will receive (20ml) (plain bupivacaine 0.25% injected in the serratus intercostal space at 6 ribs midaxillary line and (20ml) in pecto-intercostal space at 2 ribs parasternal.
  Interventions: Procedure: Ultrasound guided Thoracic Interfascial plane Block (TIFB)
- Ultrasound guided Erector Spinae plane Block (ESPB) (Experimental): Patients will receive (20ml) (plain bupivacaine 0.25% injected beneath the erector spinae muscle sheath) at the level of the fourth thoracic segment (T4).
  Interventions: Procedure: Ultrasound guided Erector Spinae plane Block (ESPB)
- General anesthesia (No Intervention): Patients will receive general anesthesia only without blocks.

INTERVENTIONS:
Procedure: Ultrasound guided Thoracic Interfascial plane Block (TIFB) — Patients of the group will be placed supine and elevate arm to the head, Serratus intercostal plane block will be with the probe in the midaxillary line, The subcutaneous tissue and serratus muscle will be identified in the superficial plane, whereas the external intercostal muscles will be identified in the intermediate plane and finally in the deep plane the ribs, pleura and lung will be identified. The needle will be advanced from caudal to cranial direction after giving 3 ml lidocaine locally. In-plane technique was used until the tip of the needle placed between the serratus anterior muscle and the external intercostals muscle a volume of 20 ml plain bupivacaine will be injected.
  Arms: Ultrasound guided Thoracic Interfascial plane Block (TIFB)
Procedure: Ultrasound guided Erector Spinae plane Block (ESPB) — The patient will be placed in setting position and a superficial (5-12 MHz) ultrasound transducer will be placed in a longitudinal orientation, 3 cm lateral to the T4 spinous process. An 8-cm 22-gauge spinal needle will be inserted in cephalic direction after giving 3 ml lidocaine locally until the needle tip hit the transverse process of T4 under ultrasound image visualization, then the needle will be withdrawn slowly to be within the interfacial plane below the erector spinae muscle, then the anesthetic mixture will be injected here. Successful injection will be evidenced by visible linear free spread (cranially and caudally) of injectate below the muscle.
  Arms: Ultrasound guided Erector Spinae plane Block (ESPB)

SUMMARY:
This study will be conducted to compare the efficacy of ultrasound guided thoracic interfascial plane block versus ultrasound guided erector spinae plane block on acute and chronic pain after modified radical mastectomy surgery.

DETAILED DESCRIPTION:
Various thoracic nerve blocks performed for pain control after breast cancer surgery provide superior analgesic effect and reduce postoperative nausea and vomiting as a result of the decreased use of opioid analgesics.

Ultrasound-guided erector spinae block (ESB) is a regional anesthesia technique; recently described by Forero et al, in management of thoracic neuropathic pain. It became popular because it is much safer and easily administered than other alternative regional techniques as paravertebral and thoracic epidural block.

ESB leads to effective postoperative analgesia when performed at T 4-5 level for breast and thoracic surgery, and T 7 level for abdominal surgeries. Spread of local anesthetic following ESB in the cephalic and caudal directions can lead to analgesia from C7 to L2-3.

There have been several reports that thoracic interfascial plane block is useful for multimodal analgesia in patients undergoing mastectomy, Thoracic interfascial plane block including pecto-intercostal fascial plane block (PIFB) and serratus intercostal fascial plane block (SIFB).

Thoracic interfascial plane block is the peripheral nerve block that targets the intercostal nerves branches distributed in the chest and axilla, Although PIFB and SIFB are thought to be relatively easy to perform there have been no reports of the simultaneous performance of the two blocks.

ELIGIBILITY:
Inclusion Criteria:

* Female patients admitted for modified radical mastectomy surgery.
* American Society of Anesthesiologists (ASA) physical activity I, II
* Aged (18 - 65) years

Exclusion Criteria:

* Patient refusal.
* Patient with neurological deficit.
* Patient with bleeding disorders (coagulopathy, thrombocytopenia anticoagulant, and antiplatelet drugs).
* Uncooperative patient.
* Infection at the block injection site.
* Patients with a history of allergy to drugs.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-10 (Estimated); Primary Completion 2022-11-24 (Estimated); Study Completion 2022-11-24 (Estimated)

PRIMARY OUTCOMES:
Total analgesics consumption in the first 24h after surgery. | 24 hours postoperative
  Total analgesic consumption (fentanyl intraoperative) and (morphine 0.05 mg / kg per dose at the first 24 h after surgery).

SECONDARY OUTCOMES:
Time to first analgesic request after surgery | 24 hours Postoperative
  Time to first analgesic request after surgery in the form of intravenous morphine in a dose (0.05 mg/kg) If VAS ≥ 4 all patient will receive paracetamol 1gm /6h.
Visual Analogue score (VAS) | 24 hours Postoperative
  Pain will be assessed after surgery over 24 hour using VAS score where (0 = no pain and 10 = severe pain) at (T 30 min, 2, 4, 6, 12, 18, 24 h), if less than 4 non-steroidal anti-inflammatory will be given (ketorolac 30mg) and if more than 4 intra venous morphine (0.05mg / kg)
Complications occurrence (hypotension, pneumothorax, bradycardia) | 24 hours Postoperative
  Adverse events as Bradycardia, hypotension, drowsiness, and dizziness) will be recorded 24 hours Postoperatively.

IPD SHARING:
Plan to Share IPD: Yes
The supporting data will be available upon a reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: one year after the end of the study